CLINICAL TRIAL: NCT05777850
Title: High-Power Short-Duration Radiofrequency Ablation in Patients With Typical Atrial Flutter
Acronym: FASD-HP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jose Luis Ibañez Criado (Other)
Responsible Party: Sponsor-Investigator, Jose Luis Ibañez Criado, Medical Doctor, Hospital General Universitario de Alicante
Organization: Hospital General Universitario de Alicante (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FASD-HP trial
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Typical Atrial Flutter; Catheter Ablation
Keywords: Typical Atrial Flutter Cavotricuspid Isthmus; Cavotricuspid Isthmus; High-Power Short-Duration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional ablation (Active Comparator): CTI ablation with electroanatomic navigation system using individual 25-40 W applications of unlimited duration until achieving in each application the minimum value of one of the currently accepted and used lesion markers: Ablation Index >500 at the anterior half of the CTI and >400 at the posterior half with de CARTO 3 system. Minimum contact force required is 5 grams. Maximum distance between applications must be 6 mm.
  Interventions: Procedure: Conventional cavotricuspid isthmus ablation
- High-power short-duration ablation (Experimental): CTI ablation with electroanatomic navigation system using individual high power (90W) short duration (4 seconds) applications in a catheters' stable position with a minimum contact force of 15-30 g at the anterior half and 10-25 g at the posterior one. Maximum distance between applications is settled at 4 mm.
  Interventions: Procedure: High-power short-duration ablation

INTERVENTIONS:
Procedure: Conventional cavotricuspid isthmus ablation — Point-by-point 25-40 W applications at the CTI of unlimited duration until achieving the pre-established Ablation Index.
  Arms: Conventional ablation
Procedure: High-power short-duration ablation — Point-by-point 90W applications at the CTI ablation during 4 seconds.
  Arms: High-power short-duration ablation

SUMMARY:
The aim of cavotricuspid isthmus (CTI) dependent flutter ablation is the bidirectional conduction block of CTI. The probability of achieving a permanent bidirectional block at the CTI depends, mainly, on the ablation energy applied and the quality of the obtained lesion. Among the factors that determine the lesion's quality those which have the bigger impact are catheter stability, contact force, power and duration of energy application and the temperature reached at depth.This is a multicenter 1:1 randomized, blinded (open for the operator) study. Two CTI ablation strategies are compared: 1) conventional treatment branch which consists of individual 25-40 W applications of unlimited duration until achieving in each application the minimum value of one of the currently accepted and used lesion markers (Ablation Index >500 at the anterior half of the CTI and >400 at the posterior half with de CARTO 3 system; 2) experimental treatment branch consistent of CTI block using individual high power (90W) short duration (4 seconds) point-by-point applications. The main objective of this study is assessing the non-inferiority of the efficacy and safety of high-power short-duration ablation in patients undergoing typical atrial flutter ablation. Secondary objectives include the comparison of total radiofrequency time, number of applications, number of steam pops, percentage of reconnections, procedure duration, pain during the procedure and time to atrial flutter recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cavotricuspid isthmus dependent flutter referred to ablation
* Patients clinically and hemodynamically stable.
* Patients who give informed consent.

Exclusion Criteria:

* Refusal to participate in the register or inability to understand the informed consent.
* Age under 18.
* Patients who have already undergone previous flutter ablation procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Safety primary outcome: incidence of procedure-related complications. | One year
  Number of procedure-related complications from the time of the ablation until the last follow-up visit.
Efficacy primary outcome: typical atrial flutter recurrence. | One year
  Incidence of typical atrial flutter recurrence during a one-year follow-up period. To be considered clinically relevant the recurrence must be documented by a full EKG made because of patients' symptoms or any typical atrial flutter detected by an EKG, 24h Holter-EKG or events-monitoring device that will be performed at least at a 6 months and 12 months follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Doctor Balmis Alicante, Alicante, A, Spain

REFERENCES:
- [Derived] Valverde Soria L, Toquero J, Brouzet T, Garcia Cano L, Garcia Barrios A, Segura Dominguez M, Hermon Ramirez GA, Ajo Ferrer R, Ajo Ferrer M, Andreu Concha CM, Arrarte Esteban V, Sanchez Barbie A, Martinez-Martinez JG, Ibanez Criado A, Ibanez Criado JL. Very high-power short-duration radiofrequency ablation in patients with typical atrial flutter: rationale and design of the FASD-HP randomized trial. J Interv Card Electrophysiol. 2025 Apr;68(3):497-503. doi: 10.1007/s10840-024-01969-7. Epub 2024 Dec 21. PMID 39708245